CLINICAL TRIAL: NCT05974891
Title: The Effect of Simulation-Based Experience on the Development of Self-Awareness and Empathic Skill in Nursing Students
Brief Title: The Effect of Simulation-Based Experience on Nursing Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gizem Kaya, Research Assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: E-74555795-050.01.04-634230
Record Dates: First submitted 2023-07-15; First posted 2023-08-03 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Empathy; Student; Self Awareness; Simulation; Education
Keywords: simulation; education; Empathic Skill; Self-awareness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Simulated group (Experimental): Pilot application will be carried out with at least 10 students. A pre-test will be applied to the experimental group. After the scales are applied, the experiment will be applied to the experimental group with the "Geriatric Medication Game" simulation.
  Students simulating the elderly patient role during this simulation will gain a better understanding of age-related health problems and how older adults feel when confronting them. After the application, debriefing, which is the last stage of the simulation training, will be done to evaluate the application. After the application and analysis session is completed, the post-test will be applied to the experimental group. A 3-week clinical practice will be planned for the students in the experimental groups in order to evaluate the continuation of the acquired skills and acquired awareness. In this application, students will be asked to care for the elderly patient and the pre-test will be repeated at the end of the application.
  Interventions: Other: Pilot application
- No Intervention: Control group (No Intervention): The control group will be pre-tested. After the scales are applied, no intervention will be made to the control group. A 3-week clinical practice will be planned for the students in the control group. In this application, students in the control group will be asked to care for the elderly patient and the scales will be repeated at the end of the application.

INTERVENTIONS:
Other: Pilot application — Pilot application will be carried out with at least 10 students. A pre-test will be applied to the experimental group. After the scales are applied, the experiment will be applied to the experimental group with the "Geriatric Medication Game" simulation.
  Students simulating the elderly patient role during this simulation will gain a better understanding of age-related health problems and how older adults feel when confronting them. After the application, debriefing, which is the last stage of the simulation training, will be done to evaluate the application. After the application and analysis session is completed, the post-test will be applied to the experimental group. A 3-week clinical practice will be planned for the students in the experimental groups in order to evaluate the continuation of the acquired skills and acquired awareness. In this application, students will be asked to care for the elderly patient and the pre-test will be repeated at the end of the application.
  Arms: Experimental: Simulated group

SUMMARY:
This research was planned as a randomized controlled experimental study to determine the effect of simulation training on the acquisition of self-awareness and empathy skills in nursing students.

DETAILED DESCRIPTION:
Simulation is defined as one of the methods that enables students to increase their knowledge and performance in an unreal, safe and risk-free environment and gain experience. Recent research involving the use of simulation in nursing education has mostly focused on the development of cognitive learning and psychomotor skills. However; A limited number of simulation studies have been found that include empirical evaluation of affective learning domains such as affective awareness, self-awareness and empathy. As well as the cognitive and psychomotor domains of nurse educators; It is very important for them to develop strategies to strengthen the affective field. It is predicted that the proportion of the elderly population in our country will increase in the coming years. With the increase in the elderly population, it is likely that there will be changes in the patient profile that nurses who are responsible for 24/7 individual care will encounter. Professional development is required to meet the needs of elderly patients. It is of great importance for nursing students who are still in the education stage to raise this awareness, to increase their self-awareness, to empathize with elderly individuals and to gain these characteristics. In this context, it is aimed to present results on the effects of the simulation scenario designed on the care of elderly individuals and the application of "Geriatric Medication Game" on the self-awareness levels and empathy skills of nursing students. Geriatric Medication Game is an aging simulation game that combines the experiences and challenges of older adults in healthcare and a structured role-playing where students assume the identity of healthcare-seeking seniors. It is designed to influence student attitudes and understanding of older adults and the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and over,
* Studying in the 4th grade,
* Having an AGNO grade point average of 1.80 and above,
* It will consist of students who agree to participate in the research.

Exclusion Criteria:

* Having a health problem that may affect the evaluation of the affective field/receiving treatment,
* Repeating courses due to failure in professional main courses,
* Refusing to participate in the research or giving up during the implementation process,
* Students who graduated from health vocational high school and received associate degree education in the field of health.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Self-Awareness In Nursing Practice Scale | It will be applied in the pre-test before recruitment. It will be applied immediately after the simulation.
  The scale, developed by Rasheed et al. (2020) to measure the self-awareness level of nurses, was conducted by Tufan and Oskay Şahin (2021), for its validity and reliability in Turkish. The original scale consists of 4 sub-dimensions and 18 items. The Turkish form of the scale consists of 4 sub-dimensions and 15 items. A 6-point Likert scale (always = 5, very often = 4, sometimes = 3, rarely = 2, very rarely =1 and never=0) is used. There is no reverse item in the scale. In the total score evaluation of the scale, the lowest total score is 0 and the highest total score is 75 (Tufan & Oskay Şahin, 2021).
Jefferson Empathy Scale for Nursing Students | It will be applied in the pre-test before recruitment. It will be applied immediately after the simulation.
  The scale developed by Hojat et al. (2001), Turkish validity-reliability study was conducted by Yanık and Saygılı (2014). The original scale consists of 20 items and 3 dimensions, but the Turkish version has 18 items. It has been reported that the 5th and 18th items in the Turkish scale were removed by the researchers because the factor load was found to be low (Yanık & Saygılı, 2014). The 18-item Turkish version of the scale, as in the original, consists of 3 dimensions: Obtaining an Empathic Perspective (9 items), Compassionate Care (7 items) and Viewing from the Patient's Perspective (2 items). The scale is 7-point Likert type and the scores that can be obtained from the Turkish form vary between 18-126. A high score indicates a high level of empathy (Yanik & Saygılı, 2014).
Kiersma-Chen Empathy Scale | It will be applied in the pre-test before recruitment. It will be applied immediately after the simulation.
  The scale developed by Kiersma et al. (2013) was adapted into Turkish by Şahin Bayındır et al. (2022). The original version of the scale consists of 2 subscales (Cognitive Empathy and Affective Empathy) and 15 items. However, in the Turkish adaptation study, two items with low item-total correlation (item 4 and item 15) were removed from the scale. The Turkish version of the scale consists of 2 sub-dimensions and 13 items. The scale is used to evaluate empathy in nursing students and simulation training. Responses to the scale items are scored on a 7-point Likert type (1=Strongly Disagree, 2=Disagree, 3=Somewhat Disagree, 4=Neither Agree Neither Disagree, 5=Agree Slightly, 6=Agree, 7=Strongly Agree) (Şahin-Bayindir et al., 2022). The internal consistency coefficient of the Cognitive Empathy Subscale of the scale, which was adapted into Turkish, was 0.78; The internal consistency of the Affective Empathy Subscale was 0.74; the internal consistency coefficient of the total scale is 0.85
Student Satisfaction and Self-Confidence Scale in Learning | It will be applied immediately after the simulation
  The scale was developed by Jeffries and Rizzolo (2006) as 13 items to measure students' simulation activity and self-confidence in learning. Answering the scale for each item; 1=Strongly Disagree, 2=Disagree, 3=Undecided, 4=Agree, 5=Strongly Agree (Franklin et al., 2014). The Turkish validity and reliability study of the scale was carried out by Unver et al. (2017) and the total number of items decreased to 12.
The Aging Simulation Experience Survey | It will be applied in the pre-test before recruitment. It will be applied immediately after the simulation.
  The scale was developed by Chen et al. (2011) to assess students' perceptions of older adults. In this quantitative scale, there are 13 items (7-point Likert type, 1=strongly disagree…7=strongly agree) to be filled before and after the activity regarding the experience of older adults in the health system and the structure of this system. Except for 2 items with negative expressions, higher scores were accepted as an indicator of greater understanding and positive perceptions (Chen et al., 2015b). In addition to 13 items, 8 items related to students' experience of navigating the health system as an older adult were reported to be filled only after the activity and student experiences related to the activity were evaluated (Chen et al., 2015a). There is no Turkish adaptation of the scale, it is being adapted into Turkish by the researcher.

SECONDARY OUTCOMES:
Self-Awareness In Nursing Practice Scale | 3 weeks after the simulation (after clinical practice)
  The scale, developed by Rasheed et al. (2020) to measure the self-awareness level of nurses, was conducted by Tufan and Oskay Şahin (2021), for its validity and reliability in Turkish. The original scale consists of 4 sub-dimensions and 18 items. The Turkish form of the scale consists of 4 sub-dimensions and 15 items. A 6-point Likert scale (always = 5, very often = 4, sometimes = 3, rarely = 2, very rarely =1 and never=0) is used. There is no reverse item in the scale. In the total score evaluation of the scale, the lowest total score is 0 and the highest total score is 75 (Tufan & Oskay Şahin, 2021).
Jefferson Empathy Scale for Nursing Students | 3 weeks after the simulation (after clinical practice)
  The scale developed by Hojat et al. (2001), Turkish validity-reliability study was conducted by Yanık and Saygılı (2014). The original scale consists of 20 items and 3 dimensions, but the Turkish version has 18 items. It has been reported that the 5th and 18th items in the Turkish scale were removed by the researchers because the factor load was found to be low (Yanık & Saygılı, 2014). The 18-item Turkish version of the scale, as in the original, consists of 3 dimensions: Obtaining an Empathic Perspective (9 items), Compassionate Care (7 items) and Viewing from the Patient's Perspective (2 items). The scale is 7-point Likert type and the scores that can be obtained from the Turkish form vary between 18-126. A high score indicates a high level of empathy (Yanik & Saygılı, 2014).
Kiersma-Chen Empathy Scale | 3 weeks after the simulation (after clinical practice)
  The scale developed by Kiersma et al. (2013) was adapted into Turkish by Şahin Bayındır et al. (2022). The original version of the scale consists of 2 subscales (Cognitive Empathy and Affective Empathy) and 15 items. However, in the Turkish adaptation study, two items with low item-total correlation (item 4 and item 15) were removed from the scale. The Turkish version of the scale consists of 2 sub-dimensions and 13 items. The scale is used to evaluate empathy in nursing students and simulation training. Responses to the scale items are scored on a 7-point Likert type (1=Strongly Disagree, 2=Disagree, 3=Somewhat Disagree, 4=Neither Agree Neither Disagree, 5=Agree Slightly, 6=Agree, 7=Strongly Agree) (Şahin-Bayindir et al., 2022). The internal consistency coefficient of the Cognitive Empathy Subscale of the scale, which was adapted into Turkish, was 0.78; The internal consistency of the Affective Empathy Subscale was 0.74; the internal consistency coefficient of the total scale is 0.85
The Aging Simulation Experience Survey | 3 weeks after the simulation (after clinical practice)
  The scale was developed by Chen et al. (2011) to assess students' perceptions of older adults. In this quantitative scale, there are 13 items (7-point Likert type, 1=strongly disagree…7=strongly agree) to be filled before and after the activity regarding the experience of older adults in the health system and the structure of this system. Except for 2 items with negative expressions, higher scores were accepted as an indicator of greater understanding and positive perceptions (Chen et al., 2015b). In addition to 13 items, 8 items related to students' experience of navigating the health system as an older adult were reported to be filled only after the activity and student experiences related to the activity were evaluated (Chen et al., 2015a). There is no Turkish adaptation of the scale, it is being adapted into Turkish by the researcher.

CONTACTS AND LOCATIONS:
Overall Officials: Funda BÜYÜKYILMAZ, PhD, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)